CLINICAL TRIAL: NCT05954572
Title: Association Between Biologic Therapy and Demodex Density in Psoriasis Patients: A Comparative Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasan Aksoy (Other)
Responsible Party: Sponsor-Investigator, Hasan Aksoy, Medical Doctor, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Other Study IDs: 939951438
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Demodicidosis
Keywords: demodicosis; demodex; psoriasis; biologic therapy; immunosupression
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- psoriasis patients receiving biologic therapy: A standardized form is going to be used to collect demographic information, and details regarding smoking and alcohol habits. Additional information regarding their treatment regimens will be recorded. Furthermore patients will be evaluated for the presence of acne, rosacea, perioral dermatitis, seborrheic dermatitis, folliculitis, blepharitis, or pityriasis folicullorum, as these conditions have been associated with an increased demodicosis. After that the standardized skin surface biopsy (SSSB) technique will be utilized to assess demodicosis.
  Interventions: Diagnostic Test: standardized skin surface biopsy (SSSB)
- treatment-naive or topically treated psoriasis patients: A standardized form is going to be used to collect demographic information, and details regarding smoking and alcohol habits. Additional information regarding their treatment regimens will be recorded. Furthermore patients will be evaluated for the presence of acne, rosacea, perioral dermatitis, seborrheic dermatitis, folliculitis, blepharitis, or pityriasis folicullorum, as these conditions have been associated with an increased demodicosis. After that the standardized skin surface biopsy (SSSB) technique will be utilized to assess demodicosis.
  Interventions: Diagnostic Test: standardized skin surface biopsy (SSSB)

INTERVENTIONS:
Diagnostic Test: standardized skin surface biopsy (SSSB) — This technique is applied in four facial localizations, including the forehead, cheeks, and nose. The surface biopsy procedure is performed as follows: one cm² area was marked on a glass slide using a fine ruler. The designated skin area for sampling is gently swabbed with a dry gauze pad to create mild irritation. Subsequently, one drop of cyanoacrylate adhesive is applied to the marked area on the glass slide. The glass slide is carefully pressed onto the skin, allowing the adhesive to adhere. After approximately one minute, the glass slide is gently lifted. The sampled area on the glass slide is examined under x10 and x40 magnification. Immersion oil is applied to enhance visualization and determine the number of Demodex parasites within the marked area. An increased demodicosis is defined as the presence of five or more Demodex parasites per square centimeter of skin.

SUMMARY:
The goal of this observational study is to investigate whether the density of Demodex mites is higher in psoriasis patients treated with biologic agents compared to treatment-naive or topically treated patients. The main question[s]it aims to answer are:

* Are Demodex mites higher in psoriasis patients treated with biologic agents?
* In which localization and with what intensity was demodicosis most common?

Participants will be assessed using standardized skin surface biopsy technique in four localization on their face .

Researchers will compare demodex intensity per cm² to see if the biologic treatments effects demodex intensity on psoriasis patients.

DETAILED DESCRIPTION:
This study employes a cross-sectional design to compare the density of Demodex mites in psoriasis patients receiving biologic therapy and those who had not yet initiated any treatment or were using topical medications only. The study is going to be conducted at Istanbul Medeniyet University Department of Dermatology between July 2023-August 2023. Ethics approval was obtained from Istanbul Medeniyet University Local Ethics Commitee (decision number:2022/0341).

A standardized form will be used to collect demographic information, and details regarding smoking and alcohol habits. Additional information regarding their treatment regimens will be recorded. Furthermore, patients will be evaluated for the presence of acne, rosacea, perioral dermatitis, seborrheic dermatitis, folliculitis, blepharitis, or pityriasis folicullorum, as these conditions have been associated with an increased Dd.

The standardized skin surface biopsy (SSSB) technique is going to be utilized to assess demodicosis. This technique will be applied in four facial localizations, including the forehead, cheeks, and nose. The surface biopsy procedure will be performed as follows: one cm² area will be marked on a glass slide using a fine ruler. The designated skin area for sampling will be gently swabbed with a dry gauze pad to create mild irritation. Subsequently, one drop of cyanoacrylate adhesive will be applied to the marked area on the glass slide. The glass slide will be carefully pressed onto the skin, allowing the adhesive to adhere. After approximately one minute, the glass slide will be gently lifted. The sampled area on the glass slide will be examined under x10 and x40 magnification. Immersion oil will be applied to enhance visualization and determine the number of Demodex parasites within the marked area. An increased Demodicosis will be defined as the presence of five or more Demodex parasites per square centimeter of skin.

Statistical analysis will be performed using Statistical Package for the Social Sciences [SPSS] v.17. Descriptive statistics will be calculated for relevant variables, including means, standard deviations, and frequencies. The independent samples t-test will be utilized to compare the Demodex densities, and the Chi-Square test will be used to compare the presence of demodicidosis between the two groups. P-values less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* pathologically or clinically diagnosed psoriasis patients receiving biologic therapy or topical therapy or treatment naive.

Exclusion Criteria:

* systemic therapy other then biologic agents including methotrexate, asitretin, cyclosporin etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: psoriasis patients aged between 18 and 70 which are diagnosed pathologically or clinically receiving biologic therapy or topical therapy .
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2023-08-14 (Estimated); Study Completion 2023-08-14 (Estimated)

PRIMARY OUTCOMES:
The standardized skin surface biopsy (SSSB) technique | 1 month
  measuring demodex intensity per cm² by applying the technique on four side of the face in both biologic therapy receiving group and control group.

CONTACTS AND LOCATIONS:
Overall Officials: hasan aksoy, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Keles H, Pancar Yuksel E, Aydin F, Senturk N. Pre-Treatment and Post-Treatment Demodex Densities in Patients under Immunosuppressive Treatments. Medicina (Kaunas). 2020 Mar 3;56(3):107. doi: 10.3390/medicina56030107. PMID 32138191
- [Result] Gazi U, Taylan-Ozkan A, Mumcuoglu KY. Immune mechanisms in human and canine demodicosis: A review. Parasite Immunol. 2019 Dec;41(12):e12673. doi: 10.1111/pim.12673. Epub 2019 Oct 8. PMID 31557333
- [Result] Marquardt-Feszler A, Cekala K, Debska-Slizien A, Imko-Walczuk B. Demodicosis among immunocompromised patients: a review. Postepy Dermatol Alergol. 2022 Oct;39(5):829-837. doi: 10.5114/ada.2022.120879. Epub 2022 Nov 9. PMID 36457664
- [Result] Forton FMN, De Maertelaer V. Which factors influence Demodex proliferation? A retrospective pilot study highlighting a possible role of subtle immune variations and sebaceous gland status. J Dermatol. 2021 Aug;48(8):1210-1220. doi: 10.1111/1346-8138.15910. Epub 2021 May 9. PMID 33969532
- [Result] Georgala S, Katoulis AC, Kylafis GD, Koumantaki-Mathioudaki E, Georgala C, Aroni K. Increased density of Demodex folliculorum and evidence of delayed hypersensitivity reaction in subjects with papulopustular rosacea. J Eur Acad Dermatol Venereol. 2001 Sep;15(5):441-4. doi: 10.1046/j.1468-3083.2001.00331.x. PMID 11763386
- [Result] Pappu R, Ramirez-Carrozzi V, Sambandam A. The interleukin-17 cytokine family: critical players in host defence and inflammatory diseases. Immunology. 2011 Sep;134(1):8-16. doi: 10.1111/j.1365-2567.2011.03465.x. Epub 2011 Jul 4. PMID 21726218